CLINICAL TRIAL: NCT04316637
Title: Early Access Program With Arimoclomol for the Treatment of Niemann-Pick Disease Type C in the US
Brief Title: Early Access Program With Arimoclomol in US Patients With NPC
Status: Available | Type: Expanded Access
Sponsor: ZevraDenmark (Industry)
Responsible Party: Sponsor
Other Study IDs: OR-ARI-EAP-NPC
Record Dates: First submitted 2020-03-18; First posted 2020-03-20 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Niemann-Pick Disease, Type C
MeSH Terms: conditions — Niemann-Pick Disease, Type C | interventions — arimoclomol

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: Arimoclomol — Participants receive prescribed arimoclomol by oral administration

SUMMARY:
NPC is a rare, relentlessly progressive, neurological disease and associated with serious morbidity and shortened life expectancy.

The purpose of this Expanded Access Program is to provide early access to arimoclomol for patients with Niemann-Pick Type C disease who, in the opinion and the clinical judgement of the treating physician, may benefit from treatment with arimoclomol.

Participants will receive treatment with arimoclomol until their doctor finds it does not help them anymore, they withdraw, or the study is stopped for any reason.

ELIGIBILITY:
Inclusion Criteria:

* The patient has a confirmed diagnosis of NPC (NPC1 or NPC2)* and at least one neurological symptom.
* The patient is two years of age or above.
* The patient is a permanent resident of US.
* If taking miglustat (Zavesca®), the patient must have been on the target dose for the past six weeks.
* If the patient is a sexually active female of child-bearing potential (post-menarche), it is agreed to use highly effective contraception during the EAP and until three weeks after the last dose of arimoclomol.
* Confirmed negative urine pregnancy test for sexually active female of child-bearing potential (post-menarche).
* All sexually active male patients with female partners of child-bearing potential (postmenarche) agree to use a condom in addition to the birth control used by their partners during treatment and until three weeks after the last dose of arimoclomol.
* If the patient has a history of seizures, the condition must be adequately controlled, i.e., the pattern of seizure activity must be stable, and the patient must be on a stable dose and regimen of antiepileptic medication during one month prior to screening.
* Patient or parent/guardian must provide written informed consent to participate in EAP.

  * In line with Patterson et al. 2017

Exclusion Criteria:

* Severe liver insufficiency.
* Renal insufficiency.
* The patient has a known or suspected allergy or intolerance to arimoclomol or its constituents.
* The patient is pregnant, planning to become pregnant (while on the EAP program) or is currently breastfeeding.
* The patient will undergo treatment with another investigational drug*, whilst participating in the program or in the 4 weeks prior to commencing treatment with arimoclomol.
* The patient is either eligible and able to participate in or is currently participating in an active interventional clinical trial within the indication.
* The patient, in the opinion of the clinician, is unable to comply with the treatment or has a medical condition that would potentially increase the risk to the patient by participation.
* The patient has a medical condition which hinders the clinician's assessment of arimoclomol safety and efficacy (e.g. certain epileptic conditions or severe cataplexy).

  * Including unlicensed product provided under an Early Access Program or equivalent compassionate use programs

Min Age: 2 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - University of Alabama Birmingham, Birmingham, Alabama
  - UCSF Benioff Children's Hospital and Research Center/ UCSF, Oakland, California
  - Children's Hospital of Orange County (CHOC), Orange, California
  - Nicklaus Children's Hospital, Miami, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Boston Childrens Hospital, Boston, Massachusetts
  - Mayo Clinic Children's Center, Rochester, Minnesota
  - New York University School of Medicine, New York, New York
  - Cincinnati Children's Hospital Medical Center (CCH), Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Dell Children's Medical Center, Austin, Texas
  - UT Health / McGovern Medical School; Division of Medical Genetics, Houston, Texas